CLINICAL TRIAL: NCT06175663
Title: Midlife Hypertension and Structural and Functional Brain MRI: Catching the First Signs of Cerebral Small Vessel Disease
Brief Title: Hyperintense: Midlife Hypertension and the Brain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL75003.091.20
Record Dates: First submitted 2023-12-06; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hypertension; Small Vessel Cerebrovascular Disease
MeSH Terms: conditions — Hypertension; Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood, EDTA plasma, citrate plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross-sectional study: To examine if there are cerebral abnormalities present following hypertension before MRI markers of SVD have manifested, we will do high-resolution 3T MRI in 100 young (18-40 years) hypertensive adults.
- Longitudinal study: In a cohort study, we will examine the effects of an increase and decrease in blood pressure on the brain. For this analysis, we will include hypertensive patients that are referred to the Radboudumc Department of Internal Medicine for a diagnostic work up on the cause(s) of their hypertension. The diagnostic procedure entails withdrawal of antihypertensives for approximately four weeks, as per the routine diagnostic protocol to allow for diagnosis of the cause of hypertension, and subsequent restart of treatment until the target blood pressure is reached (normotension). Measurements are performed just before antihypertensive medication is withdrawn (baseline), approximately four weeks after withdrawal (T=1), once patients have reached their target blood pressure and blood pressure is stable, estimated to occur within 2-4 months (T=2) and approximately 1 year after T=2 (T=3).
  Interventions: Drug: Antihypertensive medication withdrawal

INTERVENTIONS:
Drug: Antihypertensive medication withdrawal — To determine if high blood pressure is caused by an overproduction of aldosterone in the adrenal gland (i.e. primary hyperaldosteronism), the plasma aldosterone/renin ratio (ARR) can be determined. Because many common hypertensive drugs are known to interfere with this ratio, patients often have to discontinue drugs prior to screening or switch to drugs that are known not to affect ARR (i.e. doxazosin, verapamil, diltiazem, hydralazine). Drugs have to be stopped for at least four weeks (for mineralocorticoid receptor antagonists) or two weeks (for diuretics, Angiotensin Converting Enzyme (ACE) inhibitors, Angiotensin Receptor Blockers (ARBs)). This often leads to a temporary increase in blood pressure. After diagnostics are completed, medication is adjusted accordingly and blood pressure levels drop again.
  Groups: Longitudinal study

SUMMARY:
Cerebral small vessel disease (SVD) describes a set of pathologies affecting the smallest blood vessels in the brain. SVD contributes to up to a fifth of ischemic and hemorrhagic strokes en is the main vascular cause of dementia. On MRI, SVD is marked by different types of lesions, including white matter abnormalities, and small infarcts and hemorrhages. Recent studies indicate that SVD develops slowly over the years, starting presumably decades before the typical MRI lesions become apparent. High blood pressure plays an important role in the development of SVD MRI lesions. However, it remains unclear exactly how hypertension leads to vascular pathology. To gain more insight into how hypertension leads to SVD it is important to study mechanisms in individuals (largely) free of SVD, that is before midlife.

Therefore, the investigators aim to examine abnormalities in brain (micro) structure and vascular function in young patients with hypertension. Furthermore, the investigators aim to determine the effects of blood pressure increase and subsequent blood pressure reduction during a period of withdrawal and restart of blood pressure lowering drugs on brain (micro)structure and vascular function.

ELIGIBILITY:
Study 1: cross-sectional study

Inclusion Criteria:

* Age 18-40 years
* Blood pressure above 140/90 mmHg, measured within three months prior to study participation

Exclusion Criteria:

* Pre-existing cerebrovascular disease
* Pregnancy
* Contraindications for 3 T MRI
* Renal function eGFR below 30 ml/min (for Dynamic Contrast Enhanced [DCE]-MRI
* Major risk factors for acute ischemic stroke other than SVD according to the TOAST criteria, including, but not limited to, large-artery atherosclerosis, cardioembolism and vasculitis based on medical history and ultrasound of the carotids collected at baseline or any chronic disease that could lead to brain lesions mimicking SVD
* Major (neurological/psychiatric) disease (e.g. multiple sclerosis)
* Not able to give informed consent

Study 2: longitudinal study

Inclusion criteria:

* Age 18-55 years
* Undergoing diagnostic routine of temporary antihypertensive withdrawal for biochemical analysis as part of clinical work-up

Exclusion criteria:

* Pre-existing cerebrovascular disease
* Pregnancy
* Contraindications for 3 T MRI
* Renal function eGFR below 30 ml/min (for Dynamic Contrast Enhanced [DCE]-MRI
* Major risk factors for acute ischemic stroke other than SVD according to the TOAST criteria,22 including, but not limited to, large-artery atherosclerosis, cardioembolism and vasculitis based on medical history and ultrasound of the carotids collected at baseline or any chronic disease that could lead to brain lesions mimicking SVD
* Major (neurological/psychiatric) disease (e.g. multiple sclerosis)
* Not able to give informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited through the outpatient clinic of the Department of Internal Medicine of the Radboudumc and Rijnstate hospital, where they are referred to for their high blood pressure.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard neuroimaging markers of SVD, assessed using STRIVE criteria | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  This includes white matter hyperintensity volumes, lacunes, microbleeds, DWI+ positive lesions.
DCE-MRI outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Leakage rate (Ki)
DCE-MRI outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Volume fraction (Vl)
DTI outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Fractional Anisotropy (FA)
DTI outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Mean Diffusivity (MD)
DTI outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Peak Skeleton ofMean diffusivity (PSMD)
Intravoxel Incoherent Motion outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Parenchimal Diffusivity (D)
Intravoxel Incoherent Motion outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Perfusion fraction (F)
Intravoxel Incoherent Motion outcomes | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Microvascular perfusion (fD*)
Resting state fMRI | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Functional connectivity

SECONDARY OUTCOMES:
Cognition | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Cognitive functioning is assessed using a 60-min cognitive assessment covering six domains: processing speed, attention, executive functioning, verbal memory, working memory and psychomotor functioning.
Motor functioning | Baseline, four weeks after antihypertensive drug withdrawal, after 1-4 months when blood pressure is stable, 1 year later.
  Motor functioning is assessed using a 6-m walking test (in seconds) and the Timed Up & Go test (in seconds)
Blood markers | Four weeks after antihypertensive drug withdrawal and after 1-4 months when blood pressure is stable.
  This includes circulating markers of inflammation, including cytokines and chemokines, in mmol/l measured in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Frank-Erik de Leeuw, Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janssen E, de Jong JJA, Verburgt E, Ter Telgte A, van den Berg DTNA, Marques JP, Maas MC, Meijer FJA, Tuladhar AM, Riksen NP, Deinum J, Backes WH, de Leeuw FE. Higher Blood-Brain Barrier Permeability in Middle-Aged Adults With Hypertension. Hypertension. 2025 Dec;82(12):2172-2182. doi: 10.1161/HYPERTENSIONAHA.125.25290. Epub 2025 Oct 15. PMID 41091964